CLINICAL TRIAL: NCT04638790
Title: First Line Chemotherapy for Classical Hodgkin Lymphoma in Russia
Brief Title: First Line Chemotherapy for Classical Hodgkin Lymphoma in Russia (HL-Russia-1)
Acronym: HL-Russia-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-Russia-1
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hodgkin Lymphoma, Adult
Keywords: EACODD-14
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Etoposide; Cyclophosphamide; Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early favorable HL (Experimental): HL without adverse prognostic factors
  Interventions: Drug: Doxorubicin; Drug: Bleomycin; Drug: Vinblastine; Drug: Dacarbazine
- Early unfavorable HL (Experimental): Early unfavorable (stages IA-B, IIA bulky and/or extranodal lesions, age less than 50 years)
  Interventions: Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Dexamethasone
- Advanced stages HL (Experimental): (age less than 50 years)
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Dexamethasone; Drug: Dacarbazine

INTERVENTIONS:
Drug: Doxorubicin — 25 mg/m2 i.v. day 1,15 for ABVD/AVD
  Other Names: ABVD
  Arms: Early favorable HL; Early unfavorable HL
Drug: Bleomycin — 10,000 units/m2 i.v. days 1,15 for ABVD
  Other Names: ABVD
  Arms: Early favorable HL
Drug: Vinblastine — 6 mg/m2 i.v. days 1,15 for ABVD/AVD
  Other Names: ABVD
  Arms: Early favorable HL; Early unfavorable HL
Drug: Dacarbazine — 375 mg/m2 i.v. days 1,15 for ABVD/AVD
  Other Names: ABVD
  Arms: Early favorable HL; Early unfavorable HL
Drug: Etoposide — 100 mg/m2 i.v. days 1-3
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL
Drug: Doxorubicin — 50 mg/m2 i.v. day 1 for EACODD-14
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL
Drug: Cyclophosphamide — 650 mg/m2 i.v. day 1
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL
Drug: Vincristine — 1,4 mg/m2 i.v. day 8
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL
Drug: Dexamethasone — 20 mg i.v. days 1-3
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL
Drug: Dacarbazine — 375 mg/m2 i.v. day 1 for EACODD-14
  Other Names: EACODD-14
  Arms: Advanced stages HL; Early unfavorable HL

SUMMARY:
The HL-Russia-1 is a non-randomized, open-label, multicenter, phase III, 3-arm study. The primary objective is to assess efficacy, safety and progression-free survival (PFS) of different approaches (earle favorable, early unfavorable and advanced stages) to first line chemotherapy for classical Hodgkin Lymphoma (HL).

DETAILED DESCRIPTION:
The study is devoted to patients affected with Hodgkin Lymphoma in Russia.

The study aims to assess the efficacy and safety of three different approaches to first line chemotherapy for classical Hodgkin Lymphoma (HL):

1. Early favourable (stages I-IIA without unfavorable risk factors). Patients will receive two courses of standard ABVD (Adriamycin, bleomycin, vinblastine, and dacarbazine). Those with a PET-2 (positron emission tomography) negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (20 Gy). Those with a PET-2 Deauville score 4 will proceed with additional 2 ABVD courses. After that, those with a PET-4 negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (30 Gy). In case of PET-4 positive scan after 4 ABVD cycles (Deauville score 4-5) patients will be planned to perform the biopsy and in case of positive results, proceed to high-dose chemotherapy with autologous stem cell transplantation (HDT with ASCT). In case of negative results of the biopsy, they will proceed with additional 2 ABVD courses and restage again. Those with a PET-6 negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (30 Gy). In case of PET-6 positive scan (Deauville score 4-5) patients will be proceeded to HDT with ASCT.

   Those with a PET-2 Deauville score 5 after 2 ABVD courses will be planned to perform the biopsy and in case of positive results, proceed to HDT with ASCT. In case of negative results of the biopsy they will proceed with additional 2 ABVD courses and restage again. Those with a PET-4 negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (30 Gy). In case of PET-4 positive scan (Deauville score 4-5) patients will be proceeded to HDT with ASCT.
2. Early unfavorable (stages IA-B, IIA bulky and/or extranodal lesions, patients younger 50 years). Patients will receive two courses of EACODD-14 (etoposide 100 mg/m2 days 1-3, doxorubicin 50 mg/m2 day 1, cyclophosphamide 650 mg/m2 day 1, vincristine 1,4 mg/m2 day 8, dacarbazine 375 mg/m2 day 1, dexamethasone 20 mg days 1-3; cycle is repeated every 14 days). Those with a PET-2 negative scan (Deauville Score 1-3) will be deescalated to 2 courses of AVD (Adriamycin, vinblastine, and dacarbazine) and consolidative radiotherapy on initially involved site (30 Gy). Those with a PET-2-positive scan (Deauville score 4-5) will proceed with additional 2 EACODD-14 courses. After that, those with a PET-4 negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (30 Gy). In case of PET-4 positive scan after 4 EACODD-14 cycles (Deauville score 4-5) patients will proceed with additional 2 EACODD-14 courses. After that, those with a PET-6 negative scan (Deauville Score 1-3) will proceed with radiotherapy on initially involved site (30 Gy). In case of PET-6 positive scan (Deauville score 4-5) patients will be proceeded to HDT with ASCT.
3. Advanced stages (younger 50 years). Patients will receive two courses of EACODD-14. Those with a PET-2 negative scan (Deauville Score 1-3) will proceed with 4 additional courses of EACODD-14. After that, patients with residual tumor ˂ 4 cm, will stop the therapy and start the follow-up phase. Patients with residual tumor ≥ 4 cm, will undergo consolidative radiotherapy on residual tumor (30 Gy). Those with a PET-2-positive scan (Deauville score 4-5) will proceed with additional 4 additional courses of EACODD-14. After that, those with a PET-6 negative scan (Deauville Score 1-3) will proceed with radiotherapy on residual tumor ≥ 2,5 cm (30 Gy). In case of PET-6 positive scan (Deauville score 4-5) patients will be proceeded to HDT with ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical HL
* Previously untreated disease
* Age 18-5 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
* Adequate organ and marrow function as defined below: absolute neutrophil count >1,0 x109/L, platelets >75 x109/L
* Total bilirubin <2 mg/dl without a pattern consistent with Gilbert's syndrome
* Creatinine within normal institutional limits or creatinine clearance >50 mL/min/1.73 m2
* Females of childbearing must have a negative pregnancy test at medical supervision even if had been using effective contraception
* Life expectancy > 6 months
* Able to adhere to the study visit schedule and other protocol requirements
* Sign (or their legally acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Access to PET-CT (positron emission computed tomography) scans facilities

Exclusion Criteria:

* Nodular Lymphocyte Predominant HL
* Prior chemotherapy or radiation therapy
* Pregnant or lactating females
* Cardiac arrhythmia, conduction abnormalities, ischemic cardiopathy, left ventricular hypertrophy or left ventricular ejection fraction (LVEF) ≤50% at echocardiography.
* Abnormal QTc (corrected QT interval) interval prolonged (>450 msec in males; >470 msec in women)
* Uncontrolled infectious disease
* Human immunodeficiency virus (HIV) positivity or active infectious A, B or C hepatitis. HBsAg-negative patients with anti-HBc (hepatitis B core antigen) antibody and can be enrolled provided that Hepatitis B Virus (HBV)-DNA are negative and that antiviral treatment with nucleos(t)ide analogs is provided
* Uncompensated diabetes
* Refusal of adequate contraception
* Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | up to 6 months
  CR rate is defined as the proportion of patients achieving a CR after 3 months of chemotherapy (interim) and at the end of treatment
Acute Toxicity | 6 months
  The severity of the toxicities will be classified according to definitions of Common Terminology Criteria for Adverse Event (CTCAE) version 4.3. It will be determined by the incidence of severe, life- threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events (Infusion-related reactions)
Late Toxicity | 5 years
  The severity of the toxicities will be classified according to definitions of Common Terminology Criteria for Adverse Event (CTCAE) version 4.3. It will be determined by the incidence of severe, life- threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events (Infusion-related reactions)
Event-Free Survival (EFS) | 5 years
  EFS will be measured from the time from entry onto a study to any treatment failure including disease progression, or discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of new treatment lacking documented progression, or death)
Disease free survival (DFS) | 5 years
  DFS will be measured from the time of occurrence of disease-free state or attainment of a CR to disease recurrence or death as a result of lymphoma or acute toxicity of treatment

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  OS is defined as the time from entry onto the clinical trial until death as a result of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav Sarzhevskiy, PhD, Principal Investigator — State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia
Locations (2):
- Tata Memorial Hospital, Mumbai, Opd-81 Main Building, Dr. E Borges Road, Parel 400012, India
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No